CLINICAL TRIAL: NCT06598943
Title: An Adaptive, Dose-Ranging, Phase 2 Study of Eltrekibart Given Alone or in Combination With Mirikizumab for the Treatment of Adult Patients With Moderately to Severely Active Ulcerative Colitis
Brief Title: A Study of Eltrekibart and Mirikizumab in Adult Patients With Moderately to Severely Active Ulcerative Colitis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 18751; I7P-MC-DSAG (Other: Eli Lilly and Company)
Record Dates: First submitted 2024-09-13; First posted 2024-09-19 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Ulcerative Colitis; Ulcerative Colitis Chronic
Keywords: CXCR1/2 Ligand receptor antagonist; IL-23 p19 antibody; Gastrointestinal Diseases; Inflammatory Bowel Diseases; Digestive System Diseases; Colonic Diseases; Intestinal Diseases; Colitis; Colitis, Ulcerative; Anti-Inflammatory Agents; Mirikizumab; Eltrekibart; Adult; Moderate to Severe
MeSH Terms: conditions — Colitis, Ulcerative; Gastrointestinal Diseases; Inflammatory Bowel Diseases; Digestive System Diseases; Colonic Diseases; Intestinal Diseases; Colitis | interventions — mirikizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Eltrekibart + Placebo (Experimental): Participants will receive eltrekibart with placebo, eltrekibart or mirikizumab.
  Interventions: Drug: Eltrekibart; Drug: Mirikizumab; Drug: Placebo
- Mirikizumab + Placebo (Experimental): Participants will receive mirikizumab and placebo or mirikizumab.
  Interventions: Drug: Mirikizumab; Drug: Placebo
- Eltrekibart + Mirikizumab (Experimental): Participants will receive eltrekibart and mirikizumab in combination or separately as monotherapy.
  Interventions: Drug: Eltrekibart; Drug: Mirikizumab
- Placebo (Experimental): Participants will receive placebo or mirikizumab.
  Interventions: Drug: Mirikizumab; Drug: Placebo

INTERVENTIONS:
Drug: Eltrekibart — Administered
  Other Names: LY3041658
  Arms: Eltrekibart + Mirikizumab; Eltrekibart + Placebo
Drug: Mirikizumab — Administered
  Other Names: LY3074828
Drug: Placebo — Administered
  Arms: Eltrekibart + Placebo; Mirikizumab + Placebo; Placebo

SUMMARY:
The main purpose of this study is to determine the safety and efficacy of eltrekibart and mirikizumab in adult participants with moderately to severely active ulcerative colitis (UC).

DETAILED DESCRIPTION:
The study will last approximately 4-5 years. Screening is required within 35 days prior to enrollment. For each participant, the total duration of the clinical trial will be about 69 weeks including screening.

ELIGIBILITY:
Inclusion Criteria:

* Have had an established diagnosis of UC of ≥3 months in duration before baseline.
* Have moderately to severely active UC as assessed by the UC disease activity score.
* Have an inadequate response to, loss of response to, or intolerance to at least one conventional medication (including corticosteroids) or one advanced therapy (including biologics, Janus Kinase (JAK) inhibitors, or sphingosine-1-phosphate (S1P) immunomodulators).
* Are on a stable dose of certain oral UC medications (including corticosteroids).
* Must meet contraception requirements.

Exclusion Criteria:

* Have received anti-interleukin (IL)-23p19 or anti-IL-12p40 antibodies in the past.
* Have experienced a thrombotic event within 24 weeks before baseline.
* Have a current diagnosis of Crohn's Disease or certain other inflammatory gastrointestinal diseases.
* Have had certain abdominal surgeries within the past 3 months or are likely to require surgery for UC during the study.
* Have a history of certain adenomas, dysplasia's, or malignancies.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2024-10-10 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Achieving Clinical Remission | Week 12
  Percentage of Participants Achieving Clinical Remission

SECONDARY OUTCOMES:
Percentage of Participants Achieving Clinical Response | Week 12
  Percentage of Participants Achieving Clinical Response
Percentage of Participants Achieving Endoscopic Improvement | Week 12
  Percentage of Participants Achieving Endoscopic Improvement
Percentage of Participants Achieving Endoscopic Remission | Week 12
  Percentage of Participants Achieving Endoscopic Remission
Percentage of Participants Achieving Clinical Remission | Week 52
  Percentage of Participants Achieving Clinical Remission
Percentage of Participants Achieving Histologic-Endoscopic Mucosal Improvement | Week 12
  Percentage of Participants Achieving Histologic-Endoscopic Mucosal Improvement
Change From Baseline to Week 12 in Inflammatory Bowel Disease Questionnaire (IBDQ) Total Score | Baseline, Week 12
  Change From Baseline to Week 12 in IBDQ Total Score
Pharmacokinetics (PK): Trough concentrations at Steady State (Ctrough ss) of Eltrekibart | Week 12
  PK: Ctrough ss of Eltrekibart
PK: Ctrough ss of Mirikizumab | Week 12
  PK: Ctrough ss of Mirikizumab

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 8 AM - 8 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (207):
- United States (46):
  - AZ Gastro Care - Chandler, Chandler, Arizona
  - Applied Research Center of Arkansas, Little Rock, Arkansas
  - Preferred Research Partners, Little Rock, Arkansas
  - Erick Alayo Medical Corp/Gastro SB Clinic, Chula Vista, California
  - Southern California GI and Liver Centers (SCLC), Coronado, California
  - Valley View Research, Garden Grove, California
  - Om Research, LLC, Lancaster, California
  - United Medical Doctors, Los Alamitos, California
  - Clinnova Research, Orange, California
  - Prospective Research Innovations, Rancho Cucamonga, California
  - Clinical Trials Management Services, LLC, Thousand Oaks, California
  - Om Research LLC, Victorville, California
  - Peak Gastroenterology Associates, Colorado Springs, Colorado
  - Medical Research Center of Connecticut, LLC, Hamden, Connecticut
  - Novum Research, LLC, Clermont, Florida
  - I.V.A.M. Clinical & Investigational Center, LLC, Doral, Florida
  - Florida Research Institute, Lakewood Rch, Florida
  - Well Pharma Medical Research Corp., Miami, Florida
  - Reserka, Miami, Florida
  - Digestive Disease Consultants DDCJAX, Orange Park, Florida
  - Orlando Health Digestive Health Institute, Orlando, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Nodal Medical Center, Tampa, Florida
  - Research Bay,Inc., Tampa, Florida
  - GCP Clinical Research, LLC, Tampa, Florida
  - International Center for Research LLC, Tampa, Florida
  - Northwestern University, Chicago, Illinois
  - Avicenna Clinical Research - SW Gastroenterology, Oak Lawn, Illinois
  - Clinical Trials Management, LLC, Metairie, Louisiana
  - Gastroenterology Associates of Western Michigan, P.L.C., Wyoming, Michigan
  - Ellipsis Research Group, Brooklyn, New York
  - Smart Medical Research - Jackson Heights, Jackson Heights, New York
  - Pioneer Clinical Research NY, New York, New York
  - Digestive Disease Medicine of Central New York, Utica, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - GCGA Physicians, LLC dba / Gastro Health Research, Cincinnati, Ohio
  - NexGen Research, Lima, Ohio
  - Inquest Clinical Research, Baytown, Texas
  - DHR Health Gastroenterology - Edinburg, Edinburg, Texas
  - Baylor College of Medicine, Houston, Texas
  - Intergrity Research, Houston, Texas
  - Gastroenterology Research of San Antonio, San Antonio, Texas
  - Tyler Research Institute, Tyler, Texas
  - Care Access-Ogden, Ogden, Utah
  - Advanced Research Institute - South Ogden, Ogden, Utah
  - University of Washington School Medicine, Seattle, Washington
- Argentina (6):
  - CIPREC, CABA
  - Mautalen Salud e Investigacion-Centro de Osteopatías Médicas, Ciudad Autonoma de Buenos Air
  - Clínica Privada Independencia, Munro
  - CER Instituto Medico, Quilmes
  - Hospital Provincial del Centenario, Rosario
  - Centro Medico Privado de Reumatologia, SAN M. de Tucuman
- Belgium (2):
  - Chu Tivoli, La Louvière
  - CHU UCL Namur site Godinne, Yvoir
- Canada (4):
  - London Health Sciences Centre, London
  - London Digestive Disease Institute, London
  - CIUSSS de l'Est-de-l'Île-de-Montréal, Montreal
  - Montreal General Hospital, Montreal
- Colombia (3):
  - Hospital Universitario Mayor Méderi, Bogotá
  - Comité de Ética en Investigación Biomédica IPS Centro Médico Julián Coronel, Cali
  - Centro de Inmunología y Genética (CIGE), Medellín
- Croatia (6):
  - General Hospital Dr Andjelko Visic Bjelovar, Bjelovar
  - Poliklinika Borzan, Osijek
  - Special Hospital Medico, Rijeka
  - General Hospital Dr. J. Bencevic, Slavonski Brod
  - Poliklinika Solmed, Zagreb
  - University Hospital Center Zagreb, Zagreb
- Czechia (4):
  - SurGal clinic s.r.o., Brno
  - Vojenska nemocnice Brno p.o., Brno
  - Etická komise Nemocnice Slaný, Slaný
  - Etická komise Krajské nemocnice T. Bati, a. s., Zlín
- Bispebjerg Hospital, København NV, Denmark
- France (6):
  - Henri Mondor Hospital, Créteil
  - CHU De Grenoble Hopital Albert Michallon, Grenoble
  - Centre Hospitalier Departemental (CHD) Vendee, La Roche-sur-Yon
  - CHU de Nice Hopital de L'Archet, Nice
  - Hospices Civils de Lyon - Centre Hospitalier Lyon Sud -, Pierre-Bénite
  - Chu de Rouen Hopital Charles Nicolle, Rouen
- Germany (13):
  - Universitätsklinikum Augsburg, III. Medizinische Klinik Studienzentrum, Augsburg
  - Charité Campus Virchow-Klinikum, Berlin
  - Universitätsklinikum Brandenburg GmbH, Brandenburg
  - MVZ für spezialärztliche Versorgung Dr. Friedrichs GmbH, Duisburg
  - Universitätsklinikum Frankfurt Goethe-Universität, Medizinische Klinik 1, Frankfurt am Main
  - Interdisziplinäres Crohn Colitis Centrum Rhein-Main, Frankfurt am Main
  - Studiengesellschaft BSF Unternehmergesellschaft, Halle
  - HaFCED e.K. - Hamburgisches Forschungsinstitut für chronisch entzündliche Darmerkrankungen, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - Universitätsklinikum Schleswig-Holstein, Kiel
  - Klinikum Rechts der Isar der TU München, München
  - Magen-Darm-Zentrum Remscheid, Remscheid
  - Universitätsklinikum Ulm, Ulm
- Greece (7):
  - General Hospital of Athens 'Evangelismos', Athens
  - General Hospital of Athens Hippokratio, Athens
  - Sotiria Thoracic Diseases Hospital of Athens, Athens
  - Alexandra Hospital, Athens
  - PAGNI-University General Hospital of Heraklion, Heraklion
  - University Hospital of Ioannina, Ioannina
  - General Oncology Hospital of Kifissia "Agioi Anargiroi", Nea Kifissia
- Hungary (7):
  - Clinexpert Egészségügyi Szolgáltató és Kereskedelmi Kft, Budapest
  - Óbudai Egészségügyi Centrum, Budapest
  - Semmelweis University, Budapest
  - Bugát Pál Kórház, Gyöngyös
  - Clinexpert Gyöngyös Kft., Gyöngyös
  - Szegedi Tudományegyetem Szent-Györgyi Albert Klinikai Központ, Szeged
  - Fejér Megyei Szent György Egyetemi Oktató Kórház, Székesfehérvár
- Beaumont Hospital, Dublin, Dublin, Ireland
- Italy (19):
  - IRCCS - AOU di Bologna, Bologna
  - Fondazione Poliambulanza, Brescia
  - AST Pesaro Urbino - Presidio Ospedaliero Santa Croce, Fano
  - Azienda Ospedaliera Universitaria Careggi, Florence
  - A.O.U. Policlinico G. Martino, Gazzi - Messina
  - Ospedale S. Paolo, Milan
  - Azienda Ospedaliero Universitaria, Modena
  - Università di Cagliari - Presidio Policlinico Monserrato, Monserrato
  - Azienda Ospedale Università di Padova, Padua
  - Fondazione IRCCS Policlinico San Matteo, Pavia
  - Policlinico Tor Vergata, Roma
  - Ospedale Sandro Pertini, Roma
  - Policlinico Universitario Campus Bio-Medico, Rome
  - Istituto Clinico Humanitas, Rozzano
  - IRCCS Policlinico San Donato, San Donato Milanese
  - IRCCS Ospedale Casa Sollievo della Sofferenza, San Giovanni Rotondo
  - IRCCS Ospedale San Raffaele, Segrate
  - A.O.U. Citta' della Salute e della Scienza di Torino, Torino
  - SC Farmacia AO Ordine Mauriziano, Torino
- Japan (34):
  - Chiba University Hospital, Chiba
  - Fukuoka University Chikushi Hospital, Chikushino-shi
  - Saiseikai Fukuoka General Hospital, Fukuoak
  - Hachinohe City Hospital, Hachinohe-shi
  - National Hospital Organization Hirosaki General Medical Center, Hirosaki
  - Hiroshima City North Medical Center Asa Citizens Hospital, Hiroshima
  - Hiroshima University Hospital, Hiroshima
  - Tokai University Hospital, Isehara
  - Isesaki Municipal Hospital, Isesaki-shi
  - Kagoshima IBD Gastroenterology Clinic, Kagoshima
  - National Hospital Organization Kanazawa Medical Center, Kanazawa
  - Tsujinaka Hospital Kashiwanoha, Kashiwa
  - JCHO Kyushu Hospital, Kitakyushu-Shi
  - Yamanashi Prefectural Central Hospital, Kofu
  - Hoshi General Hospital Foundation, Koriyama-shi
  - Showa University Koto Toyosu Hospital, Kōtoku
  - Our Lady of the Snow St. Mary's Hospital, Kurume-shi
  - Kitasato University Kitasato Institute Hospital, Minatoku
  - Kyorin University Hospital, Mitaka
  - Iwate Medical University Hospital, Morioka
  - Nara Prefecture General Medical Center, Nara
  - Hyogo College of Medicine, Nishinomiya
  - Infusion Clinic, Osaka
  - Oita Red Cross Hospital, Ōita
  - Sapporo Higashi Tokushukai Hospital, Sapporo
  - Tokushukai Sapporo Tokushukai Hospital, Sapporo
  - Sapporo IBD Clinic, Sapporo Shi Chuo Ku
  - NTT Medical Center Tokyo, Shinagawa-KU
  - JHCO Tokyo Yamate Medical Center, Shinjuku-ku
  - Tokyo Metro Bokutoh Hospital, Sumida-ku
  - National Hospital Organization Shizuoka Medical Center, Sunto-gun
  - Toyama University Hospital, Toyama
  - Mie University Hospital, Tsu
  - Matsushima Hospital, Yokohama
- Latvia (2):
  - Liepaja Regional Hospital, Liepāja
  - Pauls Stradins Clinical Univeristy Hospital, Riga
- Poland (18):
  - ManerMed Sp z o.o. Centrum Medyczne ,Medis, Bydgoszcz
  - Centrum Medyczne Kermed Renata Bojata-Bronisz i Ewa Kowalińska Sp.j., Bydgoszcz
  - Centrum Medyczne Plejady Magdalena Celińska-Löwenhoff, Michał Żołnowski sp.k, Krakow
  - Centrum Nowoczesnych Terapii "Dobry Lekarz" sp. z o. o., Krakow
  - Topolowa Medicenter Ryszawa & Wspólnicy Sp.j., Krakow
  - Ip Clinic Sp. Z O. O., Lodz
  - Med-GASTR SP. Z O.O., SP.K., Lodz
  - Medrise Sp. z o.o, Lublin
  - Twoja Przychodnia Opolskie Centrum Medyczne, Opole
  - Twoja Przychodnia Pcm, Poznan
  - Endoskopia Sp. z.o.o., Sopot
  - Gastromed Sp. z o.o., Torun
  - H-T. Centrum Medyczne-Endoterapia, Tychy
  - NZOZ FOR MED sp. z o.o., Wadowice
  - WIP Warsaw IBD Point Profesor Kierkus, Warsaw
  - Centrum Medyczne Oporów, Wroclaw
  - VISTAMED, Wroclaw
  - Melita Medical, Wroclaw
- Romania (7):
  - Dr.Carol Davila Emergency University Central Military Hospital, Bucharest
  - S.C. Centrul Medical Medicum SRL, Bucharest
  - Colentina Clinical Hospital, Bucharest
  - Emergency University Hospital, Bucharest
  - Institutul Regional de Gastroenterologie și Hepatologie Prof. Dr. Octavian Fodor, Cluj-Napoca
  - Valahia Medical Center SRL, Ploieşti
  - S.C Centrul de Gastroenterologie Dr. Goldis S.R.L, Timișoara
- Serbia (8):
  - Clinical Center " Dr Dragisa Misovic Dedinje", Belgrade
  - Clinical Hospital Center Bezanijska Kosa, Belgrade
  - Clinical Hospital Center Zvezdara, Belgrade
  - Clinical Hospital Centre Zemun, Belgrade
  - Military Medical Academy, Belgrade
  - Clinical Center of Vojvodina, Novi Sad
  - General Hospital Pancevo, Pančevo
  - General Hospital "Djordje Joanovic", Zrenjanin
- Spain (9):
  - Centro Medico Teknon - DIGESTIVO, Barcelona
  - Hospital General Tomelloso, Ciudad Real
  - Hospital Universitario Reina Sofia Comite Etico, Córdoba
  - Hospital Universitario Juan Ramon Jimenez, Huelva
  - Hospital Universitario de Gran Canaria Doctor Negrín, Las Palmas de GC
  - Hospital Universitario La Paz, Madrid
  - Hospital Clínico Universitario de Santiago de Compostela, Santiago de Compostela
  - Hospital Universitario Virgen Macarena, Seville
  - CEIM Hospital Universitario y Politecnico la Fe, Valencia
- Turkey (Türkiye) (4):
  - Gazi University Medical Faculty Gazi Hospital, Ankara
  - Ege Universitesi Hastanesi, Izmir
  - İnönü Üniversitesi Tıp Fakültesi, Malatya
  - Mersin University Medical Faculty Hospital, Mersin

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and European Union (EU), whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/